CLINICAL TRIAL: NCT03695367
Title: A Phase 2, Open-Label Study of HTX 011 in a Multimodal Analgesic Regimen for Decreased Opioid Use Following Unilateral Open Inguinal Herniorrhaphy
Brief Title: Phase 2 Herniorrhaphy Study for Opioid Elimination
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heron Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: HTX-011-215
Record Dates: First submitted 2018-10-01; First posted 2018-10-04 (Actual); Results first posted 2021-07-02 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Postoperative Pain
Keywords: inguinal hernia; hernia; hernia surgery; postoperative pain; herniorrhaphy
MeSH Terms: conditions — Pain, Postoperative; Hernia, Inguinal; Hernia | interventions — Ibuprofen; Acetaminophen; Ketorolac

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Cohort 1: HTX-011 + MMA Regimen (Experimental): HTX-011 (bupivacaine/meloxicam), 300 mg/9 mg via instillation; non-opioid multimodal analgesic (MMA) regimen.
  Interventions: Drug: HTX-011; Device: Luer lock applicator; Device: Vial access device; Drug: Ibuprofen; Drug: Acetaminophen
- Cohort 2: HTX-011 + MMA Regimen + Ketorolac (Experimental): HTX-011 (bupivacaine/meloxicam), 300 mg/9 mg via instillation; non-opioid multimodal analgesic (MMA) regimen and IV ketorolac.
  Interventions: Drug: HTX-011; Device: Luer lock applicator; Device: Vial access device; Drug: Ibuprofen; Drug: Acetaminophen; Drug: Ketorolac

INTERVENTIONS:
Drug: HTX-011 — HTX-011 (bupivacaine/meloxicam), 300 mg/ 9 mg via instillation.
Device: Luer lock applicator — Applicator for instillation.
Device: Vial access device — Device for withdrawal of drug product.
Drug: Ibuprofen — Ibuprofen, 600 mg.
Drug: Acetaminophen — Acetaminophen, 1 g.
Drug: Ketorolac — Intraoperative IV ketorolac.
  Arms: Cohort 2: HTX-011 + MMA Regimen + Ketorolac

SUMMARY:
This is a Phase 2, open-label study in subjects undergoing unilateral open inguinal herniorrhaphy.

ELIGIBILITY:
Inclusion Criteria:

* Is scheduled to undergo a unilateral open inguinal herniorrhaphy with mesh under general anesthesia.
* Has an American Society of Anesthesiologists Physical Status of I, II, or III.
* Female subjects are eligible only if not pregnant, not lactating, not planning to become pregnant during the study, sterile; or using acceptable contraceptives.

Exclusion Criteria:

* Had any prior inguinal hernia repair except as a child (less than 6 years of age).
* Has a planned concurrent surgical procedure (eg, bilateral herniorrhaphy).
* Has a pre-existing concurrent acute or chronic painful physical/restrictive condition expected to require analgesic treatment in the postoperative period for pain.
* Has a contraindication or a known or suspected history of hypersensitivity or clinically significant idiosyncratic reaction to required study medications.
* Has known or suspected daily use of opioids for 7 or more consecutive days within the previous 6 months.
* Has taken any NSAIDs within least 10 days prior to the scheduled surgery.
* Has taken long-acting opioids within 3 days prior to the scheduled surgery.
* Has taken any opioids within 24 hours prior to the scheduled surgery.
* Has been administered bupivacaine within 5 days prior to the scheduled surgery.
* Has been administered any local anesthetic within 72 hours prior to the scheduled surgery.
* Has initiated treatment with study medications within 1 month prior to study drug administration that can impact pain control.
* Has been administered systemic steroids within 5 half-lives or 10 days prior to administration of study drug.
* Has a medical condition such that, in the opinion of the Investigator, participating in the study would pose a health risk to the subject or confound the postoperative assessments.
* As per subject history and/or medical records, has active infection or is currently undergoing treatment for Hepatitis B, Hepatitis C, or human immunodeficiency virus (HIV).
* Has uncontrolled anxiety, psychiatric, or neurological disorder.
* Had a malignancy in the last year, with the exception of nonmetastatic basal cell or squamous cell carcinoma of the skin or localized carcinoma in situ of the cervix.
* Has a known or suspected history of drug abuse, a positive drug screen on the day of surgery, or a recent history of alcohol abuse. Note: Subjects with a positive drug screen who are taking an allowed, prescribed medication that is known to result in a positive drug test (eg, amphetamine and dextroamphetamine for attention-deficit/hyperactivity disorder, benzodiazepine for anxiety disorder) may be eligible for participation in the study at the discretion of the Sponsor. Subjects taking any marijuana (medical or recreational) are not allowed to participate in the study.
* Previously participated in an HTX-011 study.
* Received an investigational product or device in a clinical trial within 30 days or within 5 elimination half-lives.
* Has undergone 3 or more surgeries within 12 months.
* Has a body mass index (BMI) >39 kg/m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Singla, MD, Study Chair — Lotus Clinical Research, LLC
Locations (5):
- United States (5):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Lotus Clinical Research, LLC, Pasadena, California
  - JBR Clinical Research, Draper, Utah
  - JBR Clinical Research, Murray, Utah
  - JBR Clinical Research, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1: HTX-011 + MMA Regimen | Cohort 2: HTX-011 + MMA Regimen + Ketorolac
Started | 33 | 30
Completed | 32 | 26
Not Completed | 1 | 4
Not completed — Missed the Day 28 visit. | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — One subject missed the Day 28 visit and one subject missed the Day 10 and Day 28 visits. | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: HTX-011 + MMA Regimen | Cohort 2: HTX-011 + MMA Regimen + Ketorolac | Total
Number analyzed (Participants) | 33 | 30 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 26 | 56
  >=65 years | 3 | 4 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (13.52) | 46.1 (14.99) | 48.7 (14.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 4
  Male | 33 | 26 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 9 | 23
  Not Hispanic or Latino | 19 | 21 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 4 | 5
  White | 30 | 26 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 33 | 30 | 63

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Receiving no Opioid Rescue
Time Frame: 72 hours
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: HTX-011 + MMA Regimen | Cohort 2: HTX-011 + MMA Regimen + Ketorolac
Number analyzed (Participants) | 33 | 30
Participants | 30 | 27

2. Secondary Outcome: Total Postoperative Opioid Consumption (in IV Morphine Milligram Equivalents [IV MME])
Time Frame: 72 hours
Population: Safety Population
Measure: Mean (Standard Deviation); unit: MME, morphine milligram equivalents
Arm/Group | Cohort 1: HTX-011 + MMA Regimen | Cohort 2: HTX-011 + MMA Regimen + Ketorolac
Number analyzed (Participants) | 33 | 30
MME, morphine milligram equivalents | 0.59 (2.141) | 1.32 (4.199)

3. Secondary Outcome: Percentge of Subjects Receiving no Opioid Rescue
Time Frame: 0-24 hours, 24-48 hours, 24-72 hours, 48-72 hours
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: HTX-011 + MMA Regimen | Cohort 2: HTX-011 + MMA Regimen + Ketorolac
Number analyzed (Participants) | 33 | 30
Participants
  0-24 hours | 30 | 27
  24-48 hours | 32 | 29
  24-72 hours | 32 | 28
  48-72 hours | 33 | 28

4. Secondary Outcome: Percentge of Subjects Receiving no Opioid Rescue
Time Frame: Day 28
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: HTX-011 + MMA Regimen | Cohort 2: HTX-011 + MMA Regimen + Ketorolac
Number analyzed (Participants) | 33 | 30
Participants | 28 | 24

5. Secondary Outcome: Percentge of Subjects in Severe Pain With Numeric Rating Scale (NRS-R; Windowed Worst Observation Carried Forward) of Pain Intensity Scores >7 on a Scale of 0-10 at Any Point. NRS-R for Pain Where 0 Equals no Pain and 10 Equals Worst Pain Imaginable.
Time Frame: 72 hours
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: HTX-011 + MMA Regimen | Cohort 2: HTX-011 + MMA Regimen + Ketorolac
Number analyzed (Participants) | 33 | 30
Participants | 5 | 6

ADVERSE EVENTS:
Time Frame: 28 Days.
Description: At each level of summarization (any event, System Organ Class, and Preferred Term), subjects reporting more than one TEAE are counted only once.
Arm/Group | Cohort 1: HTX-011 + MMA Regimen | Cohort 2: HTX-011 + MMA Regimen + Ketorolac
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/30
Other Adverse Events (participants affected / at risk) | 5/33 | 7/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: HTX-011 + MMA Regimen (N=33) | Cohort 2: HTX-011 + MMA Regimen + Ketorolac (N=30)
Headache (Nervous system disorders) | 1 | 2
Dizziness (Nervous system disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 2 | 3
Vomiting (Gastrointestinal disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/67/NCT03695367/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/67/NCT03695367/SAP_001.pdf